CLINICAL TRIAL: NCT04111757
Title: A Study to Investigate the Safety and Effectiveness of the Technolas® TENEO 317 Model 2 Excimer Laser for Laser In Situ Keratomileusis (LASIK) Surgery to Treat Myopia or Myopic Astigmatism
Brief Title: A Study With Technolas® TENEO 317 Model 2 Excimer Laser to Treat Participants With Myopia or Myopic Astigmatism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 884
Record Dates: First submitted 2019-09-30; First posted 2019-10-01 (Actual); Results first posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2022-05

CONDITIONS: Myopia; Myopic Astigmatism
Keywords: LASIK; Excimer Laser
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Technolas TENEO 317 Model 2 (Experimental): One or both eyes of participants will undergo LASIK surgery with the Technolas® TENEO 317 Model 2 (version 1.28 US software) Excimer Laser on Day 0.
  Interventions: Device: Technolas® TENEO 317 Model 2

INTERVENTIONS:
Device: Technolas® TENEO 317 Model 2 — LASIK eye surgery

SUMMARY:
The primary objective of this study is to collect safety and effectiveness data for the Technolas Teneo 317 Model 2 excimer laser for LASIK correction in participants with myopia and myopic astigmatism.

DETAILED DESCRIPTION:
Technolas TENEO 317 Model 2 excimer laser is a scanning excimer laser that operates at 193 nm ultraviolet wavelength to photoablate corneal tissue in order to achieve a refractive change. It is planned to enroll and treat up to 334 participant eyes, with an expectation that 300 study eyes will complete post-surgical follow-up for 6 months or until the point of achieved refractive stability. When a cohort of at least 300 eyes has achieved refractive stability at 6 months post-surgery, all other treated eyes that have not reached the 6-month examination may be discontinued at the Sponsor's request. Or, if 300 eyes achieve refractive stability at 9 months post-surgery, all other treated eyes that have not reached the 9-month examination may be discontinued

ELIGIBILITY:
Inclusion Criteria:

* Are 22 years of age or older.
* Have read, understood, and signed an informed consent form (ICF).
* Have demonstrated stable refraction (for example, a change of ≤0.5 D in sphere and cylinder) for a minimum of 12 months prior to surgery, verified by consecutive refractions and/or medical records or prescription history.
* Have myopic refractive error with or without astigmatism; sphere between -1.0 D and -10.00 D, cylinder between 0.0 D and -3.0 D; with a manifest refraction spherical equivalent (MRSE) between -1.0 D and -11.50 D.
* Have uncorrected distance visual acuity (UDVA) of 20/40 or worse.
* Have manifest distance best spectacle corrected visual acuity (BSCVA) of 20/25 (logarithm of the minimum angle of resolution [logMAR] 0.1) or better in an operative eye.
* Have equal to or less than 0.50 D spherical equivalent (SE) difference between cycloplegic and manifest refractions at Visit 1 (pre-operative).
* Have normal corneal topography as determined by the Investigator.
* Have discontinued use of contact lenses for at least 2 weeks (for hard or toric lenses) or 3 days (for soft contact lenses) prior to the pre-operative examination, and through the day of surgery.
* All contact lens wearers must demonstrate a stable refraction (within ±0.5 D), as determined by MRSE, on 2 consecutive examinations at least 1 week apart, in an eye to be treated and the axis of cylinder should not differ by more than 15 degrees from the baseline cycloplegic refraction.
* Have the ability to lie flat without difficulty.
* Are willing and able to comply with the schedule for all post-surgery follow-up visits.

Exclusion Criteria:

* Participants for whom the combination of their baseline corneal thickness and the planned operative parameters for the LASIK procedure would result in treatment depth less than 250 microns from corneal endothelium.
* Eyes for which the baseline manifest subjective refraction exhibits a difference greater than 0.50 D in sphere power, or a difference greater than 0.50 D in cylinder power, or a difference in cylinder axis of more than 15 degrees compared to the baseline cycloplegic subjective refraction. For manifest cylinder of less than 0.50 D, the difference in cylinder axis will not be taken into consideration.
* Participants for whom the pre-operative assessment of the cornea indicates that one or both eyes are not suitable candidates for treatment based upon the Investigator's medical judgment.
* Have evidence of retinal vascular disease.
* Have a history of or have active corneal disease or infection (for example, recurrent corneal erosion syndrome, herpes simplex, or herpes zoster keratitis) in either eye.
* Have a known sensitivity to any study medication.
* Have central corneal scars affecting visual acuity or unstable keratometry with irregular mires in an eye considered for eligibility.
* Have keratoconus, subclinical or forme fruste keratoconus, corneal dystrophy, or other corneal irregularity (for example, irregular astigmatism).
* Have visually significant or progressive cataract in an eye considered for eligibility.
* Had previous intraocular or corneal surgery in an eye considered for eligibility that might confound the outcome of the study or increase the risk to the participant.
* Use chronic medications by any administration route that may increase risk to the participant or may confound the outcome of the study, including those known to affect wound healing (for example, corticosteroids, antimetabolites).
* Are known to have acute or chronic disease or illness (for example, dry eye, cataract, glaucoma, immuno-compromised, rheumatoid arthritis, clinically significant atopic disease, acne rosacea) that would increase operative risk or may confound the results of the study.
* Are taking medications contraindicated for LASIK such as isotretinoin (Accutane) or amiodarone hydrochloride (Cordarone).
* Are known to be pregnant, lactating, or who plan to become pregnant during the course of the study.
* Have known sensitivity to medications used for standard LASIK.
* Have the presence of systemic disease likely to affect wound healing, for example, autoimmune disease, systemic connective tissue disease, diabetes, or severe atopic disease.
* Are participating in any other ophthalmic clinical trial within 30 days of screening or during this clinical trial.
* Have an ocular muscle disorder including a strabismus or nystagmus, or other disorder affecting fixation.
* Have a history of or evidence of glaucoma or are a glaucoma suspect.
* Have eyes with mesopic pupil size >7.0 millimeters (mm).
* Have a Schirmer's pre-operative test without anesthesia <4 mm/5 minutes.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2021-08-06 (Actual); Study Completion 2021-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anya Loncaric, Study Director — Bausch & Lomb Incorporated
Locations (10):
- United States (10):
  - Bausch Site 101, Newport Beach, California
  - Bausch Site 110, Blaine, Minnesota
  - Bausch Site 107, Bloomington, Minnesota
  - Bausch Site 108, Omaha, Nebraska
  - Bausch Site 106, Portsmouth, New Hampshire
  - Bausch Site 102, Amherst, New York
  - Bausch Site 104, Greensboro, North Carolina
  - Bausch Site 103, Mt. Pleasant, South Carolina
  - Bausch Site 109, Sioux Falls, South Dakota
  - Bausch Site 105, Cedar Park, Texas

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Period: Overall Study
Arm/Group | Technolas TENEO 317 Model 2
Started | 168; 333 Eyes
Completed | 168; 316 Eyes
Not Completed | 0; 17 Eyes

BASELINE CHARACTERISTICS:
Units Other Than Participants: Eyes
Arm/Group | Technolas TENEO 317 Model 2
Number analyzed (Participants) | 168
Number analyzed (Eyes) | 333
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 168
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.5 (6.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101
  Male | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19
  Not Hispanic or Latino | 149
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 18
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 140
  More than one race | 3
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 168

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eyes That Achieve MRSE Predictability Within ±0.50 Diopter (D) and ±1.00 D
Description: Predictability is defined as the difference between the attempted and achieved manifest refraction spherical equivalent (MRSE) at the time of refractive stability.
Time Frame: Assessed at Month 3 to Month 9
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Technolas TENEO 317 Model 2
Number analyzed (Participants) | 168
Number analyzed (Eyes) | 333
Eyes
  ±0.50 Diopter | 287
  ±1.00 Diopter | 302

2. Primary Outcome: Percentage of Eyes Targeted for Emmetropia That Achieve Uncorrected Distance Visual Acuity (UDVA) of 20/40 or Better
Description: Percentage of eyes targeted for emmetropia that achieve UDVA of 20/40 or better at the point at which refractive stability is reached.
Time Frame: Assessed at Month 3 to Month 9
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Technolas TENEO 317 Model 2
Number analyzed (Participants) | 168
Number analyzed (Eyes) | 333
Eyes | 304

ADVERSE EVENTS:
Time Frame: 9 months
Description: Ocular Adverse Events
Arm/Group | Technolas TENEO 317 Model 2
All-Cause Mortality (participants affected / at risk) | 0/168
Serious Adverse Events (participants affected / at risk) | 0/168
Other Adverse Events (participants affected / at risk) | 0/168

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Contact Sponsor directly for details

DOCUMENTS (2):
  • Study Protocol (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/57/NCT04111757/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-18): https://cdn.clinicaltrials.gov/large-docs/57/NCT04111757/SAP_001.pdf